CLINICAL TRIAL: NCT03113565
Title: Connected Electronic Wrist Strap for Patient Follow-up After Cardiac Surgery
Acronym: BECSuP
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/02
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Surgery; Surgery--Complications; Cardiac Disease; Physical Disability
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Count daily number of footsteps. — Using a connected electronic wristband to mainly quantify daily number of footsteps.

SUMMARY:
After cardiac surgery, patients' follow-up after discharge is a major public health issue. Since the main complications occur mostly during the first extra-hospital month, a follow-up period becomes necessary as the average duration of hospitalization tends to decrease. The resumption of normal physical activity is rarely transmitted and when complications arise, the healthcare team is most often informed late.

An electronic wristband is worn by the patient during the day, between the day of discharge from the hospital (D0) and the end of the second extra-hospital month (D60). The data recorded by the wristband include : bracelet ID, date, time and number of steps per day.

The primary objective of the study is to measure the resumption of physical activity after elective cardiac surgery. This objective will be quantified by the number of daily footsteps.

A secondary objective is to determine perioperative predictors of the physical resumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent elective cardiac surgery, regardless of indication and type of intervention.

Exclusion Criteria:

* Refuse of the patient,
* Misunderstanding of the system (electronic wristband, application) or the principle of the study (language problem, cerebral vascular sequelae),
* Pre-existing handicap that does not allow walking (not related to the cardiac pathology leading to the planned cardiac surgery).
* Patients who are unable to understand the content of the information delivered
* Pregnant women can not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent elective cardiac surgery, regardless of indication and type of intervention.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Measure the resumption of physical activity after cardiac surgery by counting the number of daily footsteps. | 2 months
  Count the number of daily footsteps

CONTACTS AND LOCATIONS:
Locations (1):
- Cmc Ambroise Pare, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ball L, Costantino F, Pelosi P. Postoperative complications of patients undergoing cardiac surgery. Curr Opin Crit Care. 2016 Aug;22(4):386-92. doi: 10.1097/MCC.0000000000000319. PMID 27309972
- [Result] Kim DH, Kim CA, Placide S, Lipsitz LA, Marcantonio ER. Preoperative Frailty Assessment and Outcomes at 6 Months or Later in Older Adults Undergoing Cardiac Surgical Procedures: A Systematic Review. Ann Intern Med. 2016 Nov 1;165(9):650-660. doi: 10.7326/M16-0652. Epub 2016 Aug 23. PMID 27548070
- [Result] Mazzeffi M, Zivot J, Buchman T, Halkos M. In-hospital mortality after cardiac surgery: patient characteristics, timing, and association with postoperative length of intensive care unit and hospital stay. Ann Thorac Surg. 2014 Apr;97(4):1220-5. doi: 10.1016/j.athoracsur.2013.10.040. Epub 2013 Dec 21. PMID 24360878
- [Result] Hulzebos EH, Smit Y, Helders PP, van Meeteren NL. Preoperative physical therapy for elective cardiac surgery patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD010118. doi: 10.1002/14651858.CD010118.pub2. PMID 23152283
- [Result] Mainini C, Rebelo PF, Bardelli R, Kopliku B, Tenconi S, Costi S, Tedeschi C, Fugazzaro S. Perioperative physical exercise interventions for patients undergoing lung cancer surgery: What is the evidence? SAGE Open Med. 2016 Oct 19;4:2050312116673855. doi: 10.1177/2050312116673855. eCollection 2016. PMID 27803808
- [Derived] Hauguel-Moreau M, Naudin C, N'Guyen L, Squara P, Rosencher J, Makowski S, Beverelli F. Smart bracelet to assess physical activity after cardiac surgery: A prospective study. PLoS One. 2020 Dec 1;15(12):e0241368. doi: 10.1371/journal.pone.0241368. eCollection 2020. PMID 33259484